CLINICAL TRIAL: NCT01986023
Title: A Randomized Controlled SMS Intervention For Improving Medication Adherence in Adult Stroke Patients
Brief Title: Improving Medication Adherence Through SMS (Short Messaging Service) in Adult Stroke Patients: a Randomised Controlled Behaviour Intervention Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Ayeesha Kamran Kamal, Associate Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: D43TW008660 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-18 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Medication Adherence; Stroke
Keywords: Stroke; Medication Adherence; SMS; Randomised
MeSH Terms: conditions — Medication Adherence; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS Short Message Service Arm plus Prescription (Experimental): Intervention is as follows: Drug reminder SMS will be sent to the participants in the intervention arm customised to their stroke prescription. These SMS will be interactive in a way that the participants will have to answer back if they have taken their medicine or not in a "Yes/No" format. Moreover behaviour change SMS will also be sent to the intervention arm twice weekly. In addition , Participants will be encouraged to take medication using a taxonomy of behavioral change intervention techniques.
  Interventions: Behavioral: SMS- Short Messaging Service
- Standard Prescriptions and Counselling (No Intervention): The usual care arm will undergo standard treatment and counselling regarding their treatment and the education regarding their medication as per standard of care. They will receive a standard written prescription and no SMS

INTERVENTIONS:
Behavioral: SMS- Short Messaging Service
  Arms: SMS Short Message Service Arm plus Prescription

SUMMARY:
The impact of medications used for secondary stroke prevention relies heavily upon patient adherence. Adherence is defined as "the extent to which a person's behavior - taking medication, following a diet, and/or executing lifestyle changes, corresponds with agreed recommendations from a health care provider." It is said that optimal adherence to medications may reduce the risk of a poor outcome by 26%.

The purpose of this study which is a non-pharmacologic behavioral study is to encourage adherence to medications in stroke survivors by tailored and specific SMS reminders. (Short Text Messages). These SMS reminders will support and assist stroke patients to take medications as prescribed and on time. We hypothesise that SMS will improve the adherence of patients to stroke medications by 2 points on the Morisky Medication Adherence Scale.

DETAILED DESCRIPTION:
Stroke remains a major cause of death and disability globally, accounting for 46.6 million disability adjusted life-years (DALYs) worldwide. More than 85% of all stroke-related deaths occur in low- and middle-income (LMI) countries. In a study from our center in Pakistan, the all-cause mortality due to stroke was 12.9% in the first year. Vascular causes in general and recurrent stroke in particular accounted for the bulk of the mortality cases. Recurrence of a stroke in Pakistan is documented to be as high as 53% in the first year, as opposed to international rates of approximately 30% in the first month. Evidence based guidelines recommend risk factor control with antiplatelet agents, anti-hypertensive medications, lipid lowering drugs and appropriate anti-diabetic therapy to reduce the risk of stroke recurrence. When taken together, the combination of an antihypertensive, statin and antiplatelet agent can reduce total stroke risk by 80%.

However, the impact of drugs used for secondary stroke prevention relies heavily upon patient adherence. Adherence is defined as "the extent to which a person's behavior - taking medication, following a diet, and/or executing lifestyle changes, corresponds with agreed recommendations from a health care provider." It is said that optimal adherence to medications may reduce the risk of a poor outcome by 26%.

The purpose of this study which is a non-pharmacologic behavioral study is to encourage adherence to medications in stroke survivors by tailored and specific SMS (Short Text Messages) reminders. These SMS reminders will support and assist stroke patients to take medications as prescribed and on time. We hypothesise that SMS will improve the adherence of patients to stroke medications by 2 points on the Morisky Medication Adherence Scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Diagnosed with stroke at least one month ago on neuroimaging (CT or MRI)
* Taking more than one drug for risk factor control
* Possessing a personal mobile phone
* Modified Rankin scores <3 (to exclude severely disabled persons)
* Able to operate sms
* Do not intend to travel outside the country in the next 2 months (because the followup period is 2 months and during this period mobile communication through sms is required)
* Give informed consent

Exclusion Criteria:

* Chronic Renal Failure (because such patients keep getting admitted often and also have several contraindications for therapy)

  * Any known malignancy
  * Enrolled in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Score | 2 months
  Subjects will undergo measurement of their medication Adherence Scores after 2 months of follow up on the Morisky Medication Adherence Questionnaire

SECONDARY OUTCOMES:
Patient Satisfaction with Intervention | 2 months
  This is a self designed tool which will measure the level of patient satisfaction in the intervention arm with the SMS intervention
Acceptability of m-Health intervention | 2 months
  This is a self designed tool which will measure the acceptability of m-Health intervention i.e. SMS among the participants in the intervention group

OTHER OUTCOMES:
SMS Reception, Quality Issues and Safety | 2 months
  1. Failure of SMS delivery at prespecified time e.g time of medication
  2. Proportion of SMS received at night i.e after 10 pm.

CONTACTS AND LOCATIONS:
Overall Officials: Ayeesha K Kamal, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Derived] Kamal AK, Shaikh Q, Pasha O, Azam I, Islam M, Memon AA, Rehman H, Akram MA, Affan M, Nazir S, Aziz S, Jan M, Andani A, Muqeet A, Ahmed B, Khoja S. A randomized controlled behavioral intervention trial to improve medication adherence in adult stroke patients with prescription tailored Short Messaging Service (SMS)-SMS4Stroke study. BMC Neurol. 2015 Oct 21;15:212. doi: 10.1186/s12883-015-0471-5. PMID 26486857
- [Derived] Kamal AK, Shaikh QN, Pasha O, Azam I, Islam M, Memon AA, Rehman H, Affan M, Nazir S, Aziz S, Jan M, Andani A, Muqeet A, Ahmed B, Khoja S. Improving medication adherence in stroke patients through Short Text Messages (SMS4Stroke)-study protocol for a randomized, controlled trial. BMC Neurol. 2015 Aug 28;15:157. doi: 10.1186/s12883-015-0413-2. PMID 26311325